CLINICAL TRIAL: NCT04376580
Title: Incidence and Implications With the Use of Nasal Cannulas During COVID-19
Brief Title: Use of the Nasal Cannula During COVID-19
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Tiva Group (Other)
Responsible Party: Principal Investigator, Carolina Frederico, Carolina Frederico A., Tiva Group
Other Study IDs: Nasal cannulas flow rate
Record Dates: First submitted 2020-04-30; First posted 2020-05-06 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: COVID 19
Keywords: Low flow nasal cannula; Anesthesia; Sedation; Regional Anesthesia
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this investigation is to determine the incidence of the use of the low flow nasal cannula in suspected or confirmed cases with Covid-19

DETAILED DESCRIPTION:
An anonymous questionnaire will be sent to a group of anesthesiologists via email which will allow to collect information about the use, or not, of the low flow nasal cannula, the type of procedure where it is used, and the type of personal protection weared.

ELIGIBILITY:
Inclusion Criteria:

* only for physicians

Exclusion Criteria:

* not physicians

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All physician
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of physician using los flow nasal cannula during COVID 19 pandemia | 1 month
  We'll send by email a link with an online quiz to a Group of physicians with questions related to the use of nasal cannula during their routine practice.

SECONDARY OUTCOMES:
Number of physician getting sick during Covid 19 pandemic | 1 month
  We'll send by email a link with an online quiz to a group of physicians with questions related to the use of nasal cannula during their routine practice, and one of the questions is about if the physician was getting sick during the Covid pandemic.

CONTACTS AND LOCATIONS:
Locations (1):
- Carolina Frederico, Buenos Aires, Buenos Aires F.D., Argentina

IPD SHARING:
Plan to Share IPD: Undecided